CLINICAL TRIAL: NCT00212329
Title: A Comparative Study Between the Cytokine Elispot, Tetramer, Immunoblot, and T Cell Proliferation Assays Using Fresh Blood Samples From Subjects With Recent Onset Type 1 Diabetes Mellitus
Brief Title: T Cell Validation Study Using Blood Samples From Subjects With Recent Onset Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: Tcell (IND) (completed)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes; Juvenile Onset Diabetes; Insulin Dependent Diabetes; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: T Cell Proliferation and Autoreactivity Assays
Procedure: Cellular Immunoblot Assays
Procedure: Tetramer Studies
Procedure: Cytokine ELISPOT

SUMMARY:
Type 1 diabetes is a condition that is caused in part by an abnormality of the immune system which occurs when T cells, which are part of the immune system, damage the insulin secreting cells (islet cells) in the pancreas. Although it is known that T cells are important mediators of the disease, progress in the development of reliable T cell assays has been modest. The purpose of this study is to learn which T cell assays are most reliable and reproducible so that the investigators can improve their understanding about how type 1 diabetes occurs.

DETAILED DESCRIPTION:
The T Cell Validation Study is designed to determine the ability of T cell assays to identify differences in responses from participants with type 1 diabetes compared to normal control subjects, and to compare four different laboratory tests which examine T cells to determine whether the measurements are quantitatively reproducible.

Antibody assays that confirm the presence of type 1 diabetes will be evaluated including: Diabetes Biochemical Autoantibody Assay (anti-GAD65, anti-ICA512, anti-insulin) and Islet Cell Autoantibody testing; genetic testing (deoxyribonucleic acid [DNA] and human leukocyte antigen [HLA]) will also be done to learn more about the T cell assays.

The following T Cell Assays will be conducted in individuals with type 1 diabetes, as well as those without type 1 diabetes:

* Cellular Immunoblot Testing
* T Cell Proliferation Assay
* Tetramer Assay
* Cytokine ELISpot Assay

ELIGIBILITY:
Inclusion Criteria:

To be eligible, individuals with type 1 diabetes must be:

* Diagnosed with type 1 diabetes within one year of first study visit
* 8-35 years of age at time of first visit
* Weigh > 40 kg (88 lbs) at time of first visit
* Individuals who will serve as control subjects who do not have type 1 diabetes cannot have a first degree or second degree relative with type 1 diabetes.

Exclusion Criteria:

Individuals must not:

* Have any major illness
* Be taking any steroid medications
* If female, should not be pregnant or breastfeeding.

Ages: 8 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay E Skyler, MD, Study Chair — Type 1 Diabetes TrialNet Study Chairman
Locations (14):
- United States (13):
  - Childrens Hospital of Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - Riley Hospital for Children, Indianapolis, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Naomi Berrie Diabetes Center, Columbia University, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- University of Bristol, Bristol, United Kingdom

REFERENCES:
- [Background] Arif S, Tree TI, Astill TP, Tremble JM, Bishop AJ, Dayan CM, Roep BO, Peakman M. Autoreactive T cell responses show proinflammatory polarization in diabetes but a regulatory phenotype in health. J Clin Invest. 2004 Feb;113(3):451-63. doi: 10.1172/JCI19585. PMID 14755342
- [Background] Bensoussan D, Passa P, Canivet J, Levy-Toledano S, Caen J. [Letter: platelet aggregation and assay of Willebrand factor during diabetes mellitus]. Nouv Presse Med. 1975 Jan 18;4(3):195. No abstract available. French. PMID 1129082
- [Background] Miyazaki I, Cheung RK, Gaedigk R, Hui MF, Van der Meulen J, Rajotte RV, Dosch HM. T cell activation and anergy to islet cell antigen in type I diabetes. J Immunol. 1995 Feb 1;154(3):1461-9. PMID 7822811
- [Background] Nagata M, Kotani R, Moriyama H, Yokono K, Roep BO, Peakman M. Detection of autoreactive T cells in type 1 diabetes using coded autoantigens and an immunoglobulin-free cytokine ELISPOT assay: report from the fourth immunology of diabetes society T cell workshop. Ann N Y Acad Sci. 2004 Dec;1037:10-5. doi: 10.1196/annals.1337.002. PMID 15699487
- [Background] Peakman M, Tree TI, Endl J, van Endert P, Atkinson MA, Roep BO; Second International Immunology of Diabetes Society Workshop for Standardization ot T-cell Assays in Type 1 Diabetes. Characterization of preparations of GAD65, proinsulin, and the islet tyrosine phosphatase IA-2 for use in detection of autoreactive T-cells in type 1 diabetes: report of phase II of the Second International Immunology of Diabetes Society Workshop for Standardization of T-cell assays in type 1 diabetes. Diabetes. 2001 Aug;50(8):1749-54. doi: 10.2337/diabetes.50.8.1749. PMID 11473034
- [Background] Reijonen H, Mallone R, Heninger AK, Laughlin EM, Kochik SA, Falk B, Kwok WW, Greenbaum C, Nepom GT. GAD65-specific CD4+ T-cells with high antigen avidity are prevalent in peripheral blood of patients with type 1 diabetes. Diabetes. 2004 Aug;53(8):1987-94. doi: 10.2337/diabetes.53.8.1987. PMID 15277377